CLINICAL TRIAL: NCT03715946
Title: Phase II Trial of Adjuvant De-Escalated Radiation + Concurrent and Adjuvant Nivolumab for Intermediate-High Risk P16+ Oropharynx Cancer
Brief Title: Adjuvant De-Escalated Radiation + Adjuvant Nivolumab for Intermediate-High Risk P16+ Oropharynx Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert L. Ferris, MD, PhD (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Robert L. Ferris, MD, PhD, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 18-034
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck; Oropharynx Squamous Cell Carcinoma
Keywords: Oropharynx Cancer; OPSCC; Nivolumab; Adjuvant therapy; De-Escalated Radiation; Squamous cell carcinoma; P16+; Head and Neck cancer; Oropharynx Squamous Cell Carcinoma; Carcinoma, Squamous Cell of Head and Neck; Transoral surgery; Radiotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms; Carcinoma, Squamous Cell; Head and Neck Neoplasms | interventions — Nivolumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiotherapy (RT) + Nivolumab Injection (Experimental): RT of 45 or 50 Gy in 25 daily fractions, 6 fractions per week. Nivolumab will be administered at 240 mg every 2 weeks during radiotherapy, and at 480 mg every 4 weeks for 6 doses after radiotherapy.
  Interventions: Drug: Nivolumab Injection; Radiation: Radiotherapy (RT)

INTERVENTIONS:
Drug: Nivolumab Injection — A fully human anti-programmed death 1 (PD-1) monoclonal antibody
  Other Names: BMS-936558
Radiation: Radiotherapy (RT) — 45-50 Gy accelerated fractionation in 25 daily fractions, 6 fractions per week

SUMMARY:
This clinical trial will evaluate a new combination of treatments for Oropharyngeal Squamous Cell cancers (OPSCC), and compare it to the current standard of care (concurrent, platinum-based chemoradiotherapy). Chemoradiotherapy is efficacious, but also associated with significant toxicities and is only suitable for patients with good performance status and without severe comorbidities. The purpose of this trial is to demonstrate equivalent oncologic outcome with fewer adverse effects and improved quality of life when compared to the standard of care.

DETAILED DESCRIPTION:
This study aims to enroll 135 patients (male and female, age 18+) who are newly diagnosed with resectable, squamous cell carcinoma or undifferentiated carcinoma of the oropharynx. Survival rate and treatment response of OPSCC varies based on HPV infection status and genotype; therefore, in this study, only patients who are HPV seropositive and have HPV type 16 will be enrolled. All patients will receive the same treatment, i.e. there is no active control group.

In this trial, patients will undergo transoral surgery followed by de-intensified adjuvant radiotherapy plus nivolumab. The radiotherapy will consist of 45 or 50 Gy (depending on tumor volume) in 25 daily fractions, 6 fractions per week. Nivolumab will be administered at a fixed dose of 240 mg over 30 minutes IV every 2 weeks during radiotherapy, and at 480 mg over 60 minutes IV every 4 weeks for 6 doses after radiotherapy. The first dose will be given prior to the first fraction of radiation (Day 1) on Day -3 (+/- 2 days), and continued every 2 weeks (+/- 2 days). Nivolumab will thus be given in weeks 2 and 4 of radiotherapy. Adjuvant nivolumab will then be given for a total of 6 additional doses after the completion of radiotherapy every 4 weeks (+/- 7 days), starting in the second or third week after the completion of radiotherapy. Doses of nivolumab may be interrupted, delayed, or discontinued depending on how well the subject tolerates the treatment. Relevant outcome measures include disease free survival (2 year post surgery); percutaneous gastronomy dependence (1-year postsurgery); acute and late toxicity; patient-reported Quality of Life measures, locoregional control and distant metastatic control.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years.
* ECOG performance status of 0 or 1.
* Patients must have newly diagnosed, histologically or cytologically confirmed squamous cell carcinoma or undifferentiated carcinoma of the oropharynx. Patients must have been determined to have resectable oropharyngeal disease. Patients with primary tumor or nodal metastasis fixed to the carotid artery, skull base or cervical spine are not eligible.
* Patients must have intermediate risk factors, as described below as determined by imaging studies (performed < 45 days prior to registration) and complete neck exam, from the skull base to the clavicles. The following imaging is required: CT scan of neck only with IV contrast or MRI. PET scan of HN and chest with IV contrasted CT correlation is encouraged prior to enrollment.

Intermediate risk features: Tobacco <10 pk-yr: T0-3 plus any one of the following: >N2b (> 5 LN's +), N2c/N3, +ENE >1 mm, or + margin (if approved by surgical chair) OR Tobacco >10 pk-yr: T0-3 plus any one of the following: any N2, N3, +ENE >1 mm, or + margin (if approved by surgical chair)

* Patients must have no evidence of distant metastases (M0)
* Patients must have biopsy-proven p16+ oropharynx cancer; the histologic evidence of invasive squamous cell carcinoma may have been obtained from the primary tumor or metastatic lymph node. It is required that patients have a positive p16 IHC (as surrogate for HPV) status from either the primary tumor or metastatic lymph node.
* Carcinoma of the oropharynx associated with HPV as determined by p16 protein expression using immunohistochemistry (IHC) performed by a CLIA approved laboratory.
* No prior radiation above the clavicles.
* Patients with a history of a curatively treated malignancy must be disease-free for at least two years except for carcinoma in situ of cervix, differentiated thyroid cancer, melanoma in-situ (if fully resected), and/or non-melanomatous skin cancer, or clinically negligible in judgement of investigator.
* Patients with the following within the last 6 months prior to registration must be evaluated by a cardiologist and / or neurologist prior to entry into the study.

  * Congestive heart failure > NYHA Class II
  * CVA / TIA
  * Unstable angina
  * Myocardial infarction (with or without ST elevation)
* Patients must have acceptable renal and hepatic function within 4 weeks prior to registration as defined below:

  * Absolute neutrophil count ≥1,500/mm3
  * Platelets ≥ 100,000/mm3
  * Total bilirubin ≤ the upper limit of normal (ULN)
  * Calculated creatinine clearance must be > 60 ml/min using the Cockcroft-Gault formula: (140-age)*wt(kg)/([Cr]*72). For women the calculation should be multiplied by 0.85
* Women must not be pregnant or breast-feeding. All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy. A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* Patient without intercurrent illness likely to interfere with protocol therapy.
* Patients must not have uncontrolled diabetes, uncontrolled infection despite antibiotics or uncontrolled hypertension within 30 days prior to registration.

Exclusion Criteria:

* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
* Treatment with any chemotherapy, radiation therapy, biologics for cancer, or investigational therapy within 30 days of first administration of study treatment (subjects with prior radiation, cytotoxic or investigational products < 4 weeks prior to treatment might be eligible after discussion between investigator and sponsor, if toxicities from the prior treatment have been resolved to Grade 1 (NCI CTCAE version 4).
* Known positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection. Subjects who test positive for HCV antibody but negative for HCV ribonucleic acid are permitted to enroll.
* Known history of testing positive for human immunodeficiency virus (HIV) and CD4 count < 200 or known acquired immunodeficiency syndrome (AIDS).
* Any Grade 4 laboratory abnormalities.
* History of allergy to study drug components.
* History of severe hypersensitivity reaction to any human monoclonal antibody.
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ferris, MD, PhD, Principal Investigator — UPMC Hillman Cancer Center
Locations (3):
- United States (3):
  - Winship Cancer Institute @ Emory University Hospital Midtown, Atlanta, Georgia
  - Providence Cancer Institute, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All trial participants
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 37
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: One-year Progression-free Survival (PFS)
Description: The probability of PFS measured from of beginning of study treatment, without local, regional or distant disease recurrence (appearance of new metastatic lesions). Measurement/determination of disease progression (recurrence) by CT and MRI, Chest X-Ray (Lesions acceptable as measurable when clearly defined and surrounded by an aerated lung), Tumor Markers, Clinical Examination (Clinically detected lesions will only be considered measurable when they are superficial (e.g., skin nodules and palpable lymph nodes). For skin lesions, documentation by color photography, including a ruler to estimate size of the lesion, Cytology and Histology (Cytologic confirmation of the neoplastic nature of any effusion that appears or worsens during treatment is required when the measurable tumor has met response or stable disease criteria, Ultrasound (Ultrasound may be used only as an alternative to clinical measurements for superficial palpable lymph nodes, subcutaneous lesions and thyroid nodules.
Time Frame: At 1 year post start of treatment
Population: All patients treated with Radiotherapy (RT) and Nivolumab with radiologic evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 40
percentage of participants | 97.50 [92.80 to 100.00]

2. Primary Outcome: Two-year Progression-free Survival (PFS)
Description: as for outcome 1
Time Frame: At 2 years post start of treatment
Population: All patients treated with Radiotherapy (RT) and Nivolumab with radiologic evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 40
percentage of participants | 90.00 [81.20 to 99.80]

3. Primary Outcome: PEG Tube Dependence
Description: Presence /absence of enteral feeding tube.
Time Frame: At 1-year post-surgery
Population: All trial participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 40
Participants
  PEG tube dependence patients | 1
  Patients not PEG tube dependent | 39

4. Secondary Outcome: Worst Grade of Adverse Events Related to Treatment
Description: Number of patients experiencing Adverse Events and Serious Adverse Events (SAE) related to study treatment per Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Time Frame: Up to 24 months
Population: All patients treated with Radiotherapy (RT) and Nivolumab.
Measure: Number; unit: participants
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 40
participants
  Grade 2 | 9
  Grade 3 | 29
  Grade 4 | 2

5. Secondary Outcome: Local Recurrence-free Survival (RFS) at One Year
Description: Probability of patients with disease growth that is not present within the area in which disease was first located. Measurement/determination of disease progression (recurrence) by CT and MRI, Chest X-Ray (Lesions acceptable as measurable when clearly defined and surrounded by an aerated lung), Tumor Markers, Clinical Examination (Clinically detected lesions will only be considered measurable when they are superficial (e.g., skin nodules and palpable lymph nodes). For skin lesions, documentation by color photography, including a ruler to estimate size of the lesion, Cytology and Histology (Cytologic confirmation of the neoplastic nature of any effusion that appears or worsens during treatment is required when the measurable tumor has met response or stable disease criteria, Ultrasound (Ultrasound may be used only as an alternative to clinical measurements for superficial palpable lymph nodes, subcutaneous lesions and thyroid nodules.
Time Frame: At 1-year post-surgery
Population: All patients treated with Radiotherapy (RT) and Nivolumab with radiologic evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 40
percentage of participants | 100.00 [100.00 to 100.00]

6. Secondary Outcome: Local Recurrence-free Survival (RFS) at Two Years
Description: as for outcome 5
Time Frame: At 2-years post-surgery
Population: All patients treated with Radiotherapy (RT) and Nivolumab with radiologic evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 40
percentage of participants | 97.50 [92.80 to 100.00]

7. Secondary Outcome: Regional Recurrence-free Survival (RFS)
Description: Probability of patients with disease growth that is not present within the anatomical region in which disease was first located. Measurement/determination of disease progression (recurrence) by CT and MRI, Chest X-Ray (Lesions acceptable as measurable when clearly defined and surrounded by an aerated lung), Tumor Markers, Clinical Examination (Clinically detected lesions will only be considered measurable when they are superficial (e.g., skin nodules and palpable lymph nodes). For skin lesions, documentation by color photography, including a ruler to estimate size of the lesion, Cytology and Histology (Cytologic confirmation of the neoplastic nature of any effusion that appears or worsens during treatment is required when the measurable tumor has met response or stable disease criteria, Ultrasound (Ultrasound may be used only as an alternative to clinical measurements for superficial palpable lymph nodes, subcutaneous lesions and thyroid nodules.
Time Frame: At one year post surgery
Population: All patients treated with Radiotherapy (RT) and Nivolumab with radiologic evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 40
percentage of participants | 100.00 [100.00 to 100.00]

8. Secondary Outcome: Regional Recurrence-free Survival (RFS)
Description: as for outcome 7
Time Frame: At two years post-surgery
Population: All patients treated with Radiotherapy (RT) and Nivolumab with radiologic evaluation.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 40
participants | 100.00 [100.00 to 100.00]

9. Secondary Outcome: Distant Recurrence-free Survival (RFS) at One Year
Description: Probability of patients with disease that has spread (metastasized) to areas farther away from where disease was first located. Measurement/determination of disease progression (recurrence) by CT and MRI, Chest X-Ray (Lesions acceptable as measurable when clearly defined and surrounded by an aerated lung), Tumor Markers, Clinical Examination (Clinically detected lesions will only be considered measurable when they are superficial (e.g., skin nodules and palpable lymph nodes). For skin lesions, documentation by color photography, including a ruler to estimate size of the lesion, Cytology and Histology (Cytologic confirmation of the neoplastic nature of any effusion that appears or worsens during treatment is required when the measurable tumor has met response or stable disease criteria, Ultrasound (Ultrasound may be used only as an alternative to clinical measurements for superficial palpable lymph nodes, subcutaneous lesions and thyroid nodules.
Time Frame: At one year post-surgery
Population: All patients treated with Radiotherapy (RT) and Nivolumab with radiologic evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 40
percentage of patients | 97.50 [92.50 to 100.00]

10. Secondary Outcome: Distant Recurrence-free Survival (RFS)
Description: Percentage of patients with disease that has spread (metastasized) to areas farther away from where disease was first located. Measurement/determination of disease progression (recurrence) by CT and MRI, Chest X-Ray (Lesions acceptable as measurable when clearly defined and surrounded by an aerated lung), Tumor Markers, Clinical Examination (Clinically detected lesions will only be considered measurable when they are superficial (e.g., skin nodules and palpable lymph nodes). For skin lesions, documentation by color photography, including a ruler to estimate size of the lesion, Cytology and Histology (Cytologic confirmation of the neoplastic nature of any effusion that appears or worsens during treatment is required when the measurable tumor has met response or stable disease criteria, Ultrasound (Ultrasound may be used only as an alternative to clinical measurements for superficial palpable lymph nodes, subcutaneous lesions and thyroid nodules.
Time Frame: At 2 years post-surgery
Population: All patients treated with Radiotherapy (RT) and Nivolumab with radiologic evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 40
percentage of patients | 92.50 [84.70 to 100.00]

11. Secondary Outcome: Overall Survival (OS) at One Year
Description: The probability of survival from the start of treatment.
Time Frame: At one year
Population: All trial participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 40
percentage of participants | 100.00 [100.00 to 100.00]

12. Secondary Outcome: Overall Survival (OS) at Two Years
Description: The probability of survival from the start of treatment.
Time Frame: At two years
Population: All trial participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 40
percentage of participants | 97.50 [92.80 to 100.00]

13. Secondary Outcome: MD Anderson Dysphagia Inventory (MDADI)
Description: The MDADI measures swallowing-related quality of life (QOL) in patients with swallowing dysfunction in a 20 - item written questionnaire. Each item is scored on a 5-point Likert scale (scoring is 5-strongly disagree, 4-disagree, 3-no opinion, 2-agree, 1-strongly agree). Subscales evaluate the patient's physical (P), emotional (E) and functional (F) perceptions of swallowing dysfunction. A composite score is generated by calculating the mean response for the 19 items (excluding the global question) making up the emotional, functional and physical subscales and multiplying the result by 20, resulting in a score ranging from 20 representing a low QOL function to 100 indicating high QOL. Higher scores indicate better perception of swallowing function.
Time Frame: At baseline
Population: All treated patients that completed the MDADI questionnaire(s) at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 39
score on a scale
  Daily Activity (one-item Global Score summary) | 3.36 (1.405)
  Composite (average across 19 items) | 74.0217 (11.16120)

14. Secondary Outcome: MD Anderson Dysphagia Inventory (MDADI)
Description: as for outcome 13
Time Frame: At 3 months after start of treatment
Population: All treated patients that completed the MDADI questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 39
score on a scale
  Daily (one-item Global Score summary) | 3.67 (1.366)
  Composite (average across 19 items) | 67.2227 (9.60136)

15. Secondary Outcome: MD Anderson Dysphagia Inventory (MDADI)
Description: as for outcome 13
Time Frame: At 6 months after start of treatment
Population: All treated patients that completed the MDADI questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 31
score on a scale
  Daily (one-item Global Score summary) | 3.80 (1.186)
  Composite (average across 19 items) | 72.8767 (13.07152)

16. Secondary Outcome: MD Anderson Dysphagia Inventory (MDADI)
Description: as for outcome 13
Time Frame: At 9 months after start of treatment
Population: All treated patients that completed the MDADI questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 2
score on a scale
  Daily (one-item Global Score summary) | 4.00 (0.000)
  Composite (average across 19 items) | 74.2105 (6.69891)

17. Secondary Outcome: MD Anderson Dysphagia Inventory (MDADI)
Description: as for outcome 13
Time Frame: At 12 months after start of treatment
Population: All treated patients that completed the MDADI questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 35
score on a scale
  Daily (one-item Global Score summary) | 3.91 (1.040)
  Composite (average across 19 items) | 76.0519 (12.03900)

18. Secondary Outcome: MD Anderson Dysphagia Inventory (MDADI)
Description: as for outcome 13
Time Frame: At 18 months after start of treatment
Population: All treated patients that completed the MDADI questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 4
score on a scale
  Daily (one-item Global Score summary) | 4.50 (.577)
  Composite (average across 19 items) | 79.8688 (16.88788)

19. Secondary Outcome: MD Anderson Dysphagia Inventory (MDADI)
Description: as for outcome 13
Time Frame: At 21 months after start of treatment
Population: All treated patients that completed the MDADI questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 2
score on a scale
  Daily (one-item Global Score summary) | 3.00 (1.414)
  Composite (average across 19 items) | 61.2871 (17.53215)

20. Secondary Outcome: MD Anderson Dysphagia Inventory (MDADI)
Description: as for outcome 13
Time Frame: At 24 months after start of treatment
Population: All treated patients that completed the MDADI questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 24
score on a scale
  Daily (one-item Global Score summary) | 3.71 (1.233)
  Composite (average across 19 items) | 74.1703 (13.44307)

21. Secondary Outcome: MD Anderson Dysphagia Inventory (MDADI)
Description: as for outcome 13
Time Frame: At 30 months after start of treatment
Population: All treated patients that completed the MDADI questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 1
score on a scale
  Daily (one-item Global Score summary) | 4.00 (NA) — Mean based on one (1) participant
  Composite (average across 19 items) | 76.8421 (NA) — Mean based on one (1) participant

22. Secondary Outcome: MD Anderson Dysphagia Inventory (MDADI) (Total - Overall Score)
Description: Total scores including all time-points for the MDADI measures swallowing-related quality of life (QOL) in patients with swallowing dysfunction in a 20 - item written questionnaire. Each item is scored on a 5-point Likert scale (scoring is 5-strongly disagree, 4-disagree, 3-no opinion, 2-agree, 1-strongly agree). Subscales evaluate the patient's physical (P), emotional (E) and functional (F) perceptions of swallowing dysfunction. A composite score is generated by calculating the mean response for the 19 items (excluding the global question) making up the emotional, functional and physical subscales and multiplying the result by 20, resulting in a score ranging from 20 representing a low QOL function to 100 indicating high QOL. Higher scores indicate better perception of swallowing function. Scores taken at month 3, 6, 12, 24 and 30 months after completion of treatment were averaged for the population and reported below.
Time Frame: Up to 30 months after start of treatment
Population: All treated patients that completed the MDADI questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 39
score on a scale
  Daily (one-item Global Score summary) | 3.70 (1.216)
  Composite (average across 19 items) | 74.0179 (12.27447)

23. Secondary Outcome: Voice Handicap Index-10 (VHI-10)
Description: The VHI-10 is a patient self-assessment instrument that quantifies patients' perception of their voice handicap. It evaluates patient's physical (P), emotional (E), and functional (F) perceptions of voice and has shown to be highly reliable for internal consistency and test-retest stability. The VHI-10 utilizes a 10-item questionnaire in which the patient circles the response that most accurately reflects his or her own experience on a linear scale (from "never" to "always"). "Always" response is scored 4 points, a "Never" response is scored 0. The remaining options are scored between 1 and 3 points. The tallied number of points for each of the subscales is computed to a total composite score. Scores for the VHI-10 range from zero-to-40, with higher scores indicating a greater voice-related handicap.
Time Frame: At baseline
Population: All treated patients that completed the VHI-10 questionnaire(s) at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 37
score on a scale | 7.2432 (8.01875)

24. Secondary Outcome: Voice Handicap Index-10 (VHI-10)
Description: as for outcome 23
Time Frame: At 3 months after completion of treatment
Population: All treated patients that completed the VHI-10 questionnaire(s) for 3-month timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 6
score on a scale | 3.8333 (4.75044)

25. Secondary Outcome: Voice Handicap Index-10 (VHI-10)
Description: as for outcome 23
Time Frame: At 6 months after completion of treatment
Population: All treated patients that completed the VHI-10 questionnaire(s) for 6-month timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 30
score on a scale | 3.7000 (4.74269)

26. Secondary Outcome: Voice Handicap Index-10 (VHI-10)
Description: as for outcome 23
Time Frame: At 9 months after completion of treatment
Population: All treated patients that completed the VHI-10 questionnaire(s) for 9-month timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 2
score on a scale | 6.0000 (5.65685)

27. Secondary Outcome: Voice Handicap Index-10 (VHI-10)
Description: as for outcome 23
Time Frame: At 12 months after completion of treatment
Population: All treated patients that completed the VHI-10 questionnaire(s) for 12-month timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 35
score on a scale | 4.5714 (5.82609)

28. Secondary Outcome: Voice Handicap Index-10 (VHI-10)
Description: as for outcome 23
Time Frame: At 18 months after completion of treatment
Population: All treated patients that completed the VHI-10 questionnaire(s) for 18-month timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 3
score on a scale | 6.0000 (6.08276)

29. Secondary Outcome: Voice Handicap Index-10 (VHI-10)
Description: as for outcome 23
Time Frame: At 21 months after completion of treatment
Population: All treated patients that completed the VHI-10 questionnaire(s) for 21-month timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 2
score on a scale | 6.0000 (1.41421)

30. Secondary Outcome: Voice Handicap Index-10 (VHI-10)
Description: as for outcome 23
Time Frame: At 24 months after completion of treatment
Population: All treated patients that completed the VHI-10 questionnaire(s) for 24-month timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 24
score on a scale | 4.1667 (5.85080)

31. Secondary Outcome: Voice Handicap Index-10 (VHI-10)
Description: as for outcome 23
Time Frame: At 30 months after completion of treatment
Population: All treated patients that completed the VHI-10 questionnaire(s) for 30-month timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 1
score on a scale | 0.0000 (NA) — Mean based on one (1) participant

32. Secondary Outcome: Voice Handicap Index-10 (VHI-10) (Total)
Description: Total scores are a mean average of time-points for the VHI-10 is a patient self-assessment instrument that quantifies patients' perception of their voice handicap. It evaluates patient's physical (P), emotional (E), and functional (F) perceptions of voice and has shown to be highly reliable for internal consistency and test-retest stability. The VHI-10 utilizes a 10-item questionnaire in which the patient circles the response that most accurately reflects his or her own experience on a linear scale (from "never" to "always"). "Always" response is scored 4 points, a "Never" response is scored 0. The remaining options are scored between 1 and 3 points. The tallied number of points for each of the subscales is computed to a total composite score. Scores for the VHI-10 range from zero-to-40, with higher scores indicating a greater voice-related handicap.
Time Frame: Calculated at 30 months after completion of treatment
Population: All treated patients that completed the VHI-10 questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 37
score on a scale | 5.0286 (6.24983)

33. Secondary Outcome: Functional Assessment of Cancer Therapy - Head and Neck Cancer (FACT-H&N) Score
Description: The FACT-H&N (version 4)17 consists of a cancer-specific questionnaire, FACT-G, in addition to 12 H&N cancer-specific items (the HN subscale). FACT-G is a 27-item measure that assesses general cancer quality of life. The FACT-G contains 4 subscales: physical, social/family, emotional, and functional well-being. Individuals are asked to indicate how true the statements are for them for the past 7 days. Subscale responses range from not at all (0), to very much (4) on a 5-point scale. Total scores range from 0 to 108, with higher scores indicating better quality of life. Total scores as mean average of the combined participant values.
Time Frame: At baseline (prior to treatment)
Population: All treated patients that completed the FACT-HN questionnaire(s) at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 38
score on a scale
  PWB | 22.5275 (5.53886)
  SWB | 25.0687 (3.18941)
  EWB | 14.5282 (1.92408)
  FWB | 19.8462 (5.46539)
  HNCS | 26.5156 (7.73295)
  FACT HN Total Score | 108.9554 (17.67586)
  FACT HN TOI | 69.2161 (16.77417)
  FACT_G | 82.1589 (10.98443)

34. Secondary Outcome: Functional Assessment of Cancer Therapy - Head and Neck Cancer (FACT-H&N) Score
Description: The FACT-H&N (version 4)17 consists of a cancer-specific questionnaire, FACT-G, in addition to 12 H&N cancer-specific items (the HN subscale). FACT-G is a 27-item measure that assesses general cancer quality of life. The FACT-G contains 4 subscales: physical, social/family, emotional, and functional well-being. Individuals are asked to indicate how true the statements are for them for the past 7 days. Subscale responses range from not at all (0), to very much (4) on a 5-point scale. Total scores range from 0 to 108, with higher scores indicating better quality of life.
Time Frame: At 3 months after start of treatment
Population: All treated patients that completed the FACT-H&N questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 7
score on a scale
  PWB | 22.2857 (4.64451)
  SWB | 23.4524 (5.08693)
  EWB | 14.7143 (1.38013)
  FWB | 19.5714 (7.56448)
  HNCS | 24.8571 (8.23465)
  FACT HN | 104.8810 (24.60323)
  FACT HN TOI | 66.7143 (19.49969)
  FACT_G | 80.0239 (17.15460)

35. Secondary Outcome: Functional Assessment of Cancer Therapy - Head and Neck Cancer (FACT-H&N) Score
Description: as for outcome 34
Time Frame: At 6 months after start of treatment
Population: All treated patients that completed the FACT-H&N questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 32
score on a scale
  PWB | 24.3438 (2.61027)
  SWB | 25.3800 (3.08092)
  EWB | 15.1562 (1.68694)
  FWB | 22.3906 (5.03013)
  HNCS | 27.4478 (6.01893)
  FACT HN | 114.7184 (14.36375)
  FACT HN TOI | 74.1822 (11.97082)
  FACT_G | 87.2706 (9.80596)

36. Secondary Outcome: Functional Assessment of Cancer Therapy - Head and Neck Cancer (FACT-H&N) Score
Description: as for outcome 34
Time Frame: At 9 months after start of treatment
Population: All treated patients that completed the FACT-H&N questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 2
score on a scale | 17.0000 (11.31371)

37. Secondary Outcome: Functional Assessment of Cancer Therapy - Head and Neck Cancer (FACT-H&N) Score
Description: as for outcome 34
Time Frame: At 12 months after start of treatment
Population: All treated patients that completed the FACT-H&N questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 35
score on a scale
  PWB | 24.1857 (4.54080)
  SWB | 25.3809 (3.77407)
  EWB | 14.5294 (1.74920)
  FWB | 22.5687 (5.73219)
  HNCS | 29.8000 (6.09146)
  FACT HN | 116.2990 (17.62760)
  FACT HN TOI | 76.4364 (14.81122)
  FACT_G | 86.6226 (12.68824)

38. Secondary Outcome: Functional Assessment of Cancer Therapy - Head and Neck Cancer (FACT-H&N) Score
Description: as for outcome 34
Time Frame: At 18 months after start of treatment
Population: All treated patients that completed the FACT-H&N questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 4
score on a scale
  PWB | 12.5000 (9.11043)
  SWB | 20.0825 (5.39882)
  EWB | 13.7500 (2.75379)
  FWB | 21.1250 (8.35040)
  HNCS | 30.5000 (9.60902)
  FACT HN | 106.9575 (31.03037)
  FACT HN TOI | 73.1250 (26.28807)
  FACT_G | 76.4575 (22.13144)

39. Secondary Outcome: Functional Assessment of Cancer Therapy - Head and Neck Cancer (FACT-H&N) Score
Description: as for outcome 34
Time Frame: At 21 months after completion of treatment
Population: All treated patients that completed the FACT-H&N questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 2
score on a scale
  PWB | 15.5000 (13.43503)
  SWB | 15.5000 (4.94975)
  EWB | 12.0000 (5.65685)
  FWB | 15.0000 (11.31371)
  HNCS | 26.0000 (4.24264)
  FACT HN | 84.0000 (39.59798)
  FACT HN TOI | 56.5000 (28.99138)
  FACT_G | 58.0000 (35.35534)

40. Secondary Outcome: Functional Assessment of Cancer Therapy - Head and Neck Cancer (FACT-H&N) Score
Description: as for outcome 34
Time Frame: At 24 months after start of treatment
Population: All treated patients that completed the FACT-H&N questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 22
score on a scale
  PWB | 23.5725 (6.02450)
  SWB | 22.3332 (5.24231)
  EWB | 14.9565 (2.34479)
  FWB | 22.3043 (6.65674)
  HNCS | 28.7317 (7.34582)
  FACT HN | 112.4083 (22.63526)
  FACT HN TOI | 75.1186 (12.41533)
  FACT_G | 83.1666 (16.99082)

41. Secondary Outcome: Functional Assessment of Cancer Therapy - Head and Neck Cancer (FACT-H&N) Score
Description: as for outcome 34
Time Frame: At 30 months after start of treatment
Population: All treated patients that completed the FACT-H&N questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 1
score on a scale
  PWB | 25.0000 (NA) — Mean based on one (1) participant
  SWB | 27.0000 (NA) — Mean based on one (1) participant
  EWB | 15.0000 (NA) — Mean based on one (1) participant
  FWB | 23.0000 (NA) — Mean based on one (1) participant
  HNCS | 32.0000 (NA) — Mean based on one (1) participant
  FACT HN | 122.0000 (NA) — Mean based on one (1) participant
  FACT HN TOI | 80.0000 (NA) — Mean based on one (1) participant
  FACT_G | 90.0000 (NA) — Mean based on one (1) participant

42. Secondary Outcome: Functional Assessment of Cancer Therapy - Head and Neck Cancer (FACT-H&N) Score (Total)
Description: Total scores as mean average of the combined timepoint values for the FACT-H&N (version 4)17 consists of a cancer-specific questionnaire, FACT-G, in addition to 12 H&N cancer-specific items (the HN subscale). FACT-G is a 27-item measure that assesses general cancer quality of life. The FACT-G contains 4 subscales: physical, social/family, emotional, and functional well-being. Individuals are asked to indicate how true the statements are for them for the past 7 days. Subscale responses range from not at all (0), to very much (4) on a 5-point scale. Total scores range from 0 to 108, with higher scores indicating better quality of life.
Time Frame: Calculated at 30 months after start of treatment
Population: All treated patients that completed the FACT-H&N questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 40
score on a scale
  PWB | 23.3432 (5.17244)
  SWB | 24.5010 (4.10237)
  EWB | 14.6476 (2.10983)
  FWB | 21.4080 (5.94202)
  HNCS | 27.9586 (6.94262)
  FACT HN | 112.0201 (19.20657)
  FACT HN TOI | 72.8599 (16.10666)
  FACT_G | 83.9290 (13.77629)

43. Secondary Outcome: MD Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN)
Description: MDASI-HN measures treatment related symptom burden in head and neck cancer patients. The 20-item MDASI measures both severity and burden of symptoms and their effect on patients' daily activities, using a numeric rating scale of 0-10. This instrument includes 13 core symptoms and 9 head and neck specific items. Higher scores indicate superior perception of function.
Time Frame: At baseline
Population: All treated patients that completed the MDASI-HN questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 40
score on a scale
  Core mean | 1.6094 (1.28258)
  Interference mean | 2.4158 (2.20166)
  HN symptoms mean | 1.2133 (1.55947)

44. Secondary Outcome: MD Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN)
Description: MDASI-HN is a 28 symptom items questionnaire of 13 general cancer-related symptoms, such as pain, fatigue and nausea; 9 HNC-related symptoms, such as problems with mucus in the mouth and difficulty in swallowing or chewing; 6 items to evaluate the effects of symptoms on daily life, including mood and enjoyment of life. Each item/subscale is rated on a 11-point scale from 0 (not at all) to 10 (as bad as you can imagine), while the items that assess the interference of symptoms on daily activities are rated from 0 (does not interfere) to 10 (interfered completely). When calculating any subscale score (arithmetic mean of items in the subscale), a majority of the subscale's items must have been responded to (ie, 7 of the 13 core symptom severity items or 4 of the 6 interference items would represent the majority of the items for the subscale). Total scores range from 0 to 280, with higher scores indicating better quality of life/lesser impairment.
Time Frame: At 3 months after start of treatment
Population: All treated patients that completed the MDASI-HN questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 6
score on a scale
  Core mean | 2.6272 (1.81460)
  Interference mean | 3.6945 (1.91017)
  HN symptoms mean | 1.1852 (1.61882)

45. Secondary Outcome: MD Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN)
Description: as for outcome 44
Time Frame: At 6 months after start of treatment
Population: All treated patients that completed the MDASI-HN questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 32
score on a scale
  Core mean | 1.4928 (.96530)
  Interference mean | 2.9615 (1.87749)
  HN symptoms mean | .6076 (.73105)

46. Secondary Outcome: MD Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN)
Description: as for outcome 44
Time Frame: At 9 months after start of treatment
Population: All treated patients that completed the MDASI-HN questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 1
score on a scale
  Core mean | 5.1538 (NA) — Mean based on one (1) participant
  Interference mean | 5.8333 (NA) — Mean based on one (1) participant
  HN symptoms mean | 3.8889 (NA) — Mean based on one (1) participant

47. Secondary Outcome: MD Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN)
Description: as for outcome 44
Time Frame: At 12 months after start of treatment
Population: All treated patients that completed the MDASI-HN questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 35
score on a scale
  Core mean | 1.7163 (1.40834)
  Interference mean | 2.5912 (1.87383)
  HN symptoms mean | .8239 (1.30055)

48. Secondary Outcome: MD Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN)
Description: as for outcome 44
Time Frame: At 18 months
Population: All treated patients that completed the MDASI-HN questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 3
score on a scale
  Core mean | 2.4615 (2.86480)
  Interference mean | 3.2222 (2.00924)
  HN symptoms mean | 1.2222 (1.92771)

49. Secondary Outcome: MD Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN)
Description: as for outcome 44
Time Frame: At 21 months after start of treatment
Population: All treated patients that completed the MDASI-HN questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 2
score on a scale
  Core mean | 3.2692 (2.66525)
  Interference mean | 3.3333 (1.41421)
  HN symptoms mean | 1.8333 (2.59272)

50. Secondary Outcome: MD Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN)
Description: as for outcome 44
Time Frame: At 24 months after start of treatment
Population: All treated patients that completed the MDASI-HN questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 24
score on a scale
  Core mean | 1.8379 (1.95695)
  Interference mean | 2.9444 (2.52938)
  HN symptoms mean | .9027 (1.61271)

51. Secondary Outcome: MD Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN)
Description: as for outcome 44
Time Frame: At 30 months after start of treatment
Population: All treated patients that completed the MDASI-HN questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 1
score on a scale
  Core mean | 1.2308 (NA) — Mean based on one (1) participant
  Interference mean | 1.0000 (NA) — Mean based on one (1) participant
  HN symptoms mean | .3333 (NA) — Mean based on one (1) participant

52. Secondary Outcome: MD Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN) (Total)
Description: Total scores as mean average of the combined timepoint values. Includes all time-points for MDASI-HN is a 28 symptom items questionnaire of 13 general cancer-related symptoms, such as pain, fatigue and nausea; 9 HNC-related symptoms, such as problems with mucus in mouth and difficulty swallowing or chewing; 6 items to evaluate the effects of symptoms on daily life, including mood and enjoyment of life. Each item/subscale is rated on a 11-point scale from 0 (not at all) to 10 (as bad as you can imagine), while the items that assess the interference of symptoms on daily activities are rated from 0 (does not interfere) to 10 (interfered completely). When calculating any subscale score (arithmetic mean of items in the subscale), a majority of the subscale's items must have been responded to (7 of the 13 core symptom severity items or 4 of the 6 interference items would represent the majority of the items for the subscale).Total scores range 0-280;higher scores mean better life quality.
Time Frame: Calculated at 30 months after start of treatment
Population: All treated patients that completed the MDASI-HN questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 40
score on a scale
  Core mean | 1.7527 (1.48249)
  Interference mean | 2.7670 (2.08132)
  HN symptoms mean | .9527 (1.38315)

53. Secondary Outcome: Modified Barium Swallow (MBS) Rating
Description: Three swallowing outcomes will be rated by the SLP conducting the MBS study and reported by research staff: 1) laryngeal penetration (yes, no); 2) aspiration (no, sensate, silent), and 3) pharyngeal residue (no, < 50%, > 50%). These have been selected as universal items generally reported by swallowing clinicians that have been shown to significantly predict pneumonia in patients with oropharyngeal cancers. Prevalence of these dysphagia endpoints will be estimated at each time point.
Time Frame: At 6 and 24 months after completion of treatment
Population: Data were not collected.
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 0

54. Secondary Outcome: Performance Status Scale (PSS-HN)
Description: The Performance Status Scale (PSS-HN) is a clinician-rated instrument consisting of 3 questions: normalcy of diet, public eating/swallowing, and understandability of speech subscales in patients with head and neck cancer. Each subscale is rated from 0 to 100, with higher scores indicating better performance.
Time Frame: At 3, 6, 12 and 24 months after completion of treatment
Population: Data were not collected.
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 0

55. Secondary Outcome: EuroQoL-5D Questionnaire
Description: EQ-5D is an instrument which evaluates the generic quality of life developed in Europe and widely used. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. A value set consists of weights that can convert each EQ-5D health profile into a value on a scale anchored at 1 (meaning full health) and 0 (meaning a state as bad as being dead). The scale allows negative values to be assigned to health states that are considered worse than dead. EQ-5D-5L index scores range from -0.59 to 1, where 1 is the best possible health state; EQ VAS scores range from 0 to 100, where 100 is the best possible health state.
Time Frame: At baseline
Population: All treated patients that completed the EQ-5D questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 40
score on a scale
  mobility | .05 (.218)
  self_care | .10 (.300)
  usual_activities | .34 (.530)
  pain_discomfort | .80 (.511)
  anxiety_depression | .39 (.586)
  Analog Scale Score | 66.450 (30.1160)

56. Secondary Outcome: EuroQoL-5D Questionnaire
Description: as for outcome 55
Time Frame: At 3 months after start of treatment
Population: All treated patients that completed the EQ-5D questionnaire(s) for 3-month timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 7
score on a scale
  mobility | .29 (.488)
  self_care | .00 (.000)
  usual_activities | .43 (.535)
  pain_discomfort | .29 (.488)
  anxiety_depression | .43 (.787)
  Analog Scale Score | 77.857 (13.4960)

57. Secondary Outcome: EuroQoL-5D Questionnaire
Description: as for outcome 55
Time Frame: At 6 months after start of treatment
Population: All treated patients that completed the EQ-5D questionnaire(s) at the 6-month timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 31
score on a scale
  mobility | .03 (.183)
  self_care | .03 (.180)
  usual_activities | .16 (.374)
  pain_discomfort | .39 (.495)
  anxiety_depression | .10 (.301)
  Analog Scale Score | 75.017 (28.8526)

58. Secondary Outcome: EuroQoL-5D Questionnaire
Description: as for outcome 55
Time Frame: At 9 months after start of treatment
Population: All treated patients that completed the EQ-5D questionnaire(s) at the 9-month timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 2
score on a scale
  mobility | .00 (.000)
  self_care | .50 (.707)
  usual_activities | 1.00 (1.414)
  pain_discomfort | 1.00 (1.414)
  anxiety_depression | .50 (.707)
  Analog Scale Score | 62.500 (45.9619)

59. Secondary Outcome: EuroQoL-5D Questionnaire
Description: as for outcome 55
Time Frame: At 12 months after start of treatment
Population: All treated patients that completed the EQ-5D questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 35
score on a scale
  mobility | .10 (.292)
  self_care | .14 (.430)
  usual_activities | .30 (.571)
  pain_discomfort | .51 (.612)
  anxiety_depression | .16 (.359)
  Analog Scale Score | 75.348 (27.3823)

60. Secondary Outcome: EuroQoL-5D Questionnaire
Description: as for outcome 55
Time Frame: At 18 months after start of treatment
Population: All treated patients that completed the EQ-5D questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 4
score on a scale
  mobility | .00 (.000)
  self_care | .25 (.500)
  usual_activities | .50 (1.000)
  pain_discomfort | .50 (1.000)
  anxiety_depression | .25 (.500)
  Analog Scale Score | 75.000 (17.3205)

61. Secondary Outcome: EuroQoL-5D Questionnaire
Description: as for outcome 55
Time Frame: At 21 months after start of treatment
Population: All treated patients that completed the EQ-5D questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 2
score on a scale
  usual_activities | 1.00 (1.414)
  pain_discomfort | 1.00 (1.414)
  anxiety_depression | .50 (.707)
  Analog Scale Score | 55.000 (21.2132)

62. Secondary Outcome: EuroQoL-5D Questionnaire
Description: as for outcome 55
Time Frame: At 24 months after start of treatment
Population: All treated patients that completed the EQ-5D questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 23
score on a scale
  mobility | .13 (.344)
  self_care | .18 (.501)
  usual_activities | .30 (.559)
  pain_discomfort | .43 (.662)
  anxiety_depression | .26 (.449)
  Analog Scale Score | 73.891 (25.4058)

63. Secondary Outcome: EuroQoL-5D Questionnaire
Description: as for outcome 55
Time Frame: At 30 months after start of treatment
Population: All treated patients that completed the EQ-5D questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 1
score on a scale
  mobility | .00 (NA) — Mean based on one (1) participant
  self_care | .00 (NA) — Mean based on one (1) participant
  usual_activities | .00 (NA) — Mean based on one (1) participant
  pain_discomfort | .00 (NA) — Mean based on one (1) participant
  anxiety_depression | .00 (NA) — Mean based on one (1) participant
  Analog Scale Score | 85.000 (NA) — Mean based on one (1) participant

64. Secondary Outcome: EuroQoL-5D Questionnaire (Total)
Description: Total scores as mean average of the combined timepoint values for the EQ-5D is an instrument which evaluates the generic quality of life developed in Europe and widely used. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. A value set consists of weights that can convert each EQ-5D health profile into a value on a scale anchored at 1 (meaning full health) and 0 (meaning a state as bad as being dead). The scale allows negative values to be assigned to health states that are considered worse than dead. EQ-5D-5L index scores range from -0.59 to 1, where 1 is the best possible health state; EQ VAS scores range from 0 to 100, where 100 is the best possible health state.
Time Frame: Calculated at 30 months after start of treatment
Population: All treated patients that completed the EQ-5D questionnaire(s).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
Number analyzed (Participants) | 40
score on a scale
  mobility | .08 (.269)
  self_care | .11 (.357)
  usual_activities | .31 (.558)
  pain_discomfort | .55 (.611)
  anxiety_depression | .25 (.478)
  Analog Scale Score | 72.250 (27.3426)

65. Other Pre Specified Outcome: Tumor TP53 Mutation
Description: Determination of tumor TP53 mutation as measured in serum and/or tissue samples. The presence of TP53 mutations results in a protein that is less able to control cell proliferation as it is unable to trigger apoptosis in cells with damaged DNA.
Time Frame: At baseline prior to treatment; Up to 5 years
Reporting Status: Not Posted

66. Other Pre Specified Outcome: Determination of Tumor Genomics
Description: Determination of tumor genomics, measured in serum and/or tissue samples. This measure will explore the of DNA sequence and gene expression differences in tumor cells and gene abnormalities may that drive the drives disease growth.
Time Frame: At baseline prior to treatment; Up to 5 years
Reporting Status: Not Posted

67. Other Pre Specified Outcome: Presence of Plasma Cytokines
Description: Determination of cytokines present in plasma samples. The presence of cytokines in tissues can associated positively or negatively in the development of disease.
Time Frame: At baseline prior to treatment; Up to 5 years
Reporting Status: Not Posted

68. Other Pre Specified Outcome: Antigen-specific Immune Response to Human Papillomavirus (HPV)
Description: Determination of antigen-specific cellular immune response to Human papillomavirus (HPV) measured in serum and/or tissue samples.
Time Frame: At baseline prior to treatment; Up to 5 years
Reporting Status: Not Posted

69. Other Pre Specified Outcome: Determination of Oral Human Papillomavirus (HPV) DNA
Description: Determination of oral HPV DNA present/measured in oral tissue samples.
Time Frame: At baseline prior to treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 24 months post treatment
Description: Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Arm/Group | Radiotherapy (RT) + Nivolumab Injection
All-Cause Mortality (participants affected / at risk) | 2/40
Serious Adverse Events (participants affected / at risk) | 4/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiotherapy (RT) + Nivolumab Injection (N=40)
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Multi-organ failure (General disorders) | 1
Abdominal infection (Infections and infestations) | 1
Bone infection (Infections and infestations) | 1
Pre-Vertebral Abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Subphrenic Abscess (Infections and infestations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Aspiration (Musculoskeletal and connective tissue disorders) | 1
Respiratory failure (Musculoskeletal and connective tissue disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiotherapy (RT) + Nivolumab Injection (N=40)
Anemia (Blood and lymphatic system disorders) | 12
serum amylase increased (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Carotid Stenosis (Cardiac disorders) | 1
cholesterol high (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 8
Sinus tachycardia (Cardiac disorders) | 6
Ear pain (Ear and labyrinth disorders) | 4
erythema r ear (Ear and labyrinth disorders) | 1
External ear pain (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 2
hypoacusis (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 4
Hypothyroidism (Endocrine disorders) | 12
Blurred vision (Eye disorders) | 3
Flashing lights (Eye disorders) | 1
Floaters (Eye disorders) | 1
light flashing (Eye disorders) | 1
macular Degeneration (Eye disorders) | 1
Watering eyes (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 14
Dental caries (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 35
Dysphagia (Gastrointestinal disorders) | 29
Esophagitis (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Gagging (thick secretions) (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 17
Gum swelling (Gastrointestinal disorders) | 1
Heartburn (Gastrointestinal disorders) | 1
Increase in gag reflex and oral mucus expectoration (Gastrointestinal disorders) | 1
mouth ulceration (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 30
Nausea (Gastrointestinal disorders) | 22
Oral dysesthesia (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 19
oral radionecrosis (Gastrointestinal disorders) | 1
Oral Ulceration (Gastrointestinal disorders) | 1
oral ulcers (Gastrointestinal disorders) | 1
Salivary duct inflammation (Gastrointestinal disorders) | 16
tongue swelling (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 6
Chills (General disorders) | 2
dysgeusia (General disorders) | 1
Edema face (General disorders) | 1
Facial pain (General disorders) | 2
Fatigue (General disorders) | 35
Fever (General disorders) | 2
Flu like symptoms (General disorders) | 1
Gait disturbance (General disorders) | 1
generalized weakness (General disorders) | 1
internal cheek pain, bilateral (General disorders) | 1
Localized edema (General disorders) | 1
Malaise (General disorders) | 2
Neck edema (General disorders) | 5
night sweats (General disorders) | 1
Pain (General disorders) | 7
pain, arms & back (General disorders) | 1
Right Ear Pain (General disorders) | 1
submandibular lymphedema (General disorders) | 1
Throat Pain general (General disorders) | 3
thrush general (General disorders) | 1
fatty liver (Hepatobiliary disorders) | 1
Hypoimmunoglobulinemia (Immune system disorders) | 1
bronchitis (Infections and infestations) | 1
cold (Infections and infestations) | 1
cold, runny nose (Infections and infestations) | 1
folliculitis (Infections and infestations) | 1
Mucosal infection (Infections and infestations) | 4
oral infection (Infections and infestations) | 1
oral mucositis (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
shingles (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Thrush (Infections and infestations) | 9
Urinary tract infection (Infections and infestations) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 20
scar band formation, R base of tongue (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 4
BPH Inv (Investigations) | 1
Cholesterol high (Investigations) | 9
Creatinine increased (Investigations) | 2
facial pain (Investigations) | 1
gout inv (Investigations) | 1
Hemoglobin increased (Investigations) | 2
hyperlipidemia inv (Investigations) | 2
indigestion (Investigations) | 1
intermittent head fog & fuzziness (Investigations) | 1
Lipase increased (Investigations) | 5
Low testosterone (Investigations) | 1
Lymphocyte count decreased (Investigations) | 29
neck pain (Investigations) | 1
Neutrophil count decreased (Investigations) | 7
Serum amylase increased (Investigations) | 8
shoulder pain inv (Investigations) | 1
splenomegaly (Investigations) | 1
swelling midde finger (Investigations) | 1
TSH increase (Investigations) | 1
Vitamin D deficiency inv (Investigations) | 1
Weight loss (Investigations) | 31
White blood cell decreased (Investigations) | 15
white blood cells increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 15
Dehydration (Metabolism and nutrition disorders) | 2
Diabetes - Type II (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 9
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyperlipidemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 18
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone growth: R inner mandible (Musculoskeletal and connective tissue disorders) | 1
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Gout (Musculoskeletal and connective tissue disorders) | 2
Hernia (Musculoskeletal and connective tissue disorders) | 1
jaw muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Jaw Pain (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 3
Left jaw pain (Musculoskeletal and connective tissue disorders) | 1
Left neck numbness (Musculoskeletal and connective tissue disorders) | 1
Limited range of motion (Musculoskeletal and connective tissue disorders) | 1
lumbar disc disease (Musculoskeletal and connective tissue disorders) | 1
Mass scapula (Musculoskeletal and connective tissue disorders) | 1
muscle soreness, neck (Musculoskeletal and connective tissue disorders) | 1
muscle spasm (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 16
neck stiffness (Musculoskeletal and connective tissue disorders) | 4
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
R shoulder impairment (Musculoskeletal and connective tissue disorders) | 1
radiation fibrosis (Musculoskeletal and connective tissue disorders) | 3
right jaw pain (Musculoskeletal and connective tissue disorders) | 1
Right Shoulder Pain (Musculoskeletal and connective tissue disorders) | 2
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 2
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 4
ageusia (Nervous system disorders) | 1
Chronic migraine without aura (Nervous system disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 6
Dysesthesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 33
Dysphasia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 7
oral paresthesia (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 8
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischemic attacks (Nervous system disorders) | 1
Trigeminal nerve disorder (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 12
Claustrophobia (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 7
Insomnia (Psychiatric disorders) | 8
Mild Mood disorder (Psychiatric disorders) | 1
Tobacco Abuse (Psychiatric disorders) | 1
BPH (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Renal insufficiency (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
urolithiasis (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Premature menopause (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 8
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 6
chest Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
gagging (Respiratory, thoracic and mediastinal disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 5
increased mucous (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Post Nasal Drip (Respiratory, thoracic and mediastinal disorders) | 1
postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
runny nose (Respiratory, thoracic and mediastinal disorders) | 1
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 7
Sore throat (Respiratory, thoracic and mediastinal disorders) | 25
Thick Mucous (Respiratory, thoracic and mediastinal disorders) | 1
thick phlegm (Respiratory, thoracic and mediastinal disorders) | 2
Throat Pain (Respiratory, thoracic and mediastinal disorders) | 1
Upper lobe and lower lobe groundglass opacities (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1
cold sore (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 8
eczema (Skin and subcutaneous tissue disorders) | 1
erythema (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Erythema, right neck (Skin and subcutaneous tissue disorders) | 1
Formication (Skin and subcutaneous tissue disorders) | 1
goosebumps, cold, skin crawling (Skin and subcutaneous tissue disorders) | 1
goosebumps, skin crawling (Skin and subcutaneous tissue disorders) | 1
lip ulcer (Skin and subcutaneous tissue disorders) | 1
neck nodule (Skin and subcutaneous tissue disorders) | 1
oral ulcer, cold sore (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 10
psoriasis (Skin and subcutaneous tissue disorders) | 1
psoriasis, forehead (Skin and subcutaneous tissue disorders) | 1
radiation dermatitis (Skin and subcutaneous tissue disorders) | 3
rash (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
right neck pain, tightness (Skin and subcutaneous tissue disorders) | 1
right neck, left back, bleeding skin spots (Skin and subcutaneous tissue disorders) | 1
Right palate and tonsillar fossa erythema and ulcerations (Skin and subcutaneous tissue disorders) | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
skin erythema (Skin and subcutaneous tissue disorders) | 2
Aortic Aneurysm (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Hypertension (Vascular disorders) | 24
Hypotension (Vascular disorders) | 4
Lymphedema (Vascular disorders) | 15
Thromboembolic event (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/46/NCT03715946/Prot_SAP_001.pdf